CLINICAL TRIAL: NCT03639961
Title: The Effect of Integrated Health System Leading, Managing and Governing for Result Model Towards Institutional Delivery Among Staff of Health Facilities in Northwest Ethiopia
Brief Title: The Effect of Integrated Leading, Managing and Governing for Result Model Towards Institutional Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bahir Dar University (Other)
Responsible Party: Principal Investigator, Yeshambel Agumas Ambelie, Lecturer, Bahir Dar University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 090/18-04
Record Dates: First submitted 2018-07-09; First posted 2018-08-21 (Actual); Last update posted 2019-06-06 (Actual); Status verified 2019-06

CONDITIONS: Leadership
Keywords: Integrated; leading; managing; governing; practices
MeSH Terms: interventions — Disease Management

STUDY DESIGN:
Intervention Model Description: The integrated health system leading, managing and governing for results model is constructed from: leading practices, managing practice, and governing practices; moderating factors ; health services performance, and sustainable health outcomes and impact aligned with national health goals and Sustainable Development Goals (SDGs).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Staff of facilities for intervention (Experimental): Intervention: Participants have been trained two times in six months period with integrated leading, managing and governing for results model.
  Interventions: Behavioral: Integrated leading, managing and governing for results model
- Staff of facilities for control (Active Comparator): Intervention: Participants have been trained two times in six months period with traditional model.
  Interventions: Behavioral: Traditional model

INTERVENTIONS:
Behavioral: Integrated leading, managing and governing for results model — Integrated leading, managing and governing for results model is an intervention launched to improve institutional delivery.
  Arms: Staff of facilities for intervention
Behavioral: Traditional model — Traditional model is a health service delivery model already in place in the government health system.
  Arms: Staff of facilities for control

SUMMARY:
The need for leading people, managing work, and governing organizations never changed over the civilization paths of society. However, people in every pole of the globe observe: over-led and under-managed, over-managed and under-governed, and even out of these organizations. These disparities have remained worse in the health system of developing countries like Ethiopia.

To date, Ethiopia put a goal of ending preventable child and maternal death, in achieving universal healthcare by 2035. Nevertheless, the investment on integrated leadership, management and governance is limited.

Therefore, this study hypothesize that institutional delivery are expressively linked with integrated health system leading, managing and governing for results model among health facilities staff in northwest Ethiopia?

DETAILED DESCRIPTION:
The investment on integrated health system leading, managing and governing for result model narrow down health system gaps.

The need to integrate these three distinct, but not hostile paths is that mostly: leading is people oriented process, managing is task oriented process and governing is organization oriented path.

Moreover, these paths are reflected even in a single person, task, or organization. Thus, testing and implementing integrated model is cost effective.

ELIGIBILITY:
Inclusion Criteria:

* All staff nominated by the respective districts that have been selected, but not deployed yet, for integrated health system leadership, management and governance for intervention by Amhara regional health office in the study setting have been included.

Exclusion Criteria:

* No exclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 418 (Actual)
Dates: Start 2018-04-10 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
Institutional delivery | Up to six months
  Increased institutional delivery. These have been assessed by institutional delivery follow up checklist. To declare that integrated leading, managing and governing for result model has an effect on institutional delivery improvement, on which it could be increased at least by 15%.

SECONDARY OUTCOMES:
Habit of institutional delivery | two weeks
  Improvement on habit of institutional delivery has been explored from key informants, by key informant guideline. The explored data will be analyzed thematically, using the Qualitative Data Analysis (QDA) miner 4 software.

CONTACTS AND LOCATIONS:
Overall Officials: G D Alene, PhD, Study Director — Bahir Dar University
Locations (1):
- North Achefer district, Līben, Amhara, Ethiopia

IPD SHARING:
Plan to Share IPD: Yes
The IPD will be shared up on the intervention study report has been published.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: From October 2019 to June 2020
Access Criteria: For any humanistic purposes

REFERENCES:
- [Derived] Silva JAM, Mininel VA, Fernandes Agreli H, Peduzzi M, Harrison R, Xyrichis A. Collective leadership to improve professional practice, healthcare outcomes and staff well-being. Cochrane Database Syst Rev. 2022 Oct 10;10(10):CD013850. doi: 10.1002/14651858.CD013850.pub2. PMID 36214207